CLINICAL TRIAL: NCT02577055
Title: Fertility After Myomectomy Versus Uterine Artery Embolization for Symptomatic Uterine Fibroids
Acronym: Lune2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P140311
Record Dates: First submitted 2015-07-20; First posted 2015-10-16 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Leiomyoma
Keywords: Leiomyoma; Uterine Artery Embolization; Surgery; childbearing age; Fertility; Noninferiority trial
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- myomectomy (Active Comparator): Women will be treated with surgical removal of all fibroids, either by laparoscopic or abdominal route
  Interventions: Procedure: myomectomy
- embolisation (Experimental): Women will be treated with fertility sparing uterine arteries embolization (i..e. with ultra thin catheter, and particles' diameter > 500µm)
  Interventions: Procedure: embolisation

INTERVENTIONS:
Procedure: myomectomy — Surgical ablation of all fibroids
  Arms: myomectomy
Procedure: embolisation — Embolisation of the peri-myoma vascular network, with non-resorbable particles of >500 µm diameter, using an ultra thin catheter introduced through the vascular network up to the uterine arteries under radioscopic control.
  Other Names: Fertility sparing ultra selective uterine artery embolization
  Arms: embolisation

SUMMARY:
Purpose of this study:

To establish the superiority of myomectomy versus Uterine Artery Embolization, in women with multiple symptomatic fibroids and no other infertility factor, seeking to conceive.

DETAILED DESCRIPTION:
Background:

The use of uterine artery embolization (UAE) to treat symptomatic fibroids in women seeking future fertility remains a matter of debate, because of possible adverse effects on ovarian reserve and embryo implantation. In women with associated infertility factors, not eligible for myomectomy, poor fertility was obtained after UAE. On the other hand, fertility of women eligible for surgical myomectomy, deciding to have a UAE, compares favourably with the fertility obtained after myomectomy.

Study design:

Eligible women will be explored to pull out any other infertility factors such as:

* tubal factors (no hydrosalpinx at MRI, tubal permeability assessed by hysterosalpingography and/or negative serology of for Chlamydia)
* Endometriosis (clinical history and examination, MRI)
* Ovarian factors (normal AMH dosage, and Antral follicular count)
* Male factors (normal spermogram of the Partner if possible)

Women will be treated with fertility sparing ultra selective uterine artery embolization, or surgical removal of multiple myomas.

A six months convalescence/cicatrisation period will be respected, then women will be allowed to intend to conceive.

Several elements will be prospectively followed:

* Spontaneous pregnancy from 6 months to 18 months after treatment
* Pregnancy outcomes
* Symptoms and quality of live with UFS-QoL and WHQ questionnaires, at 3, 6, 12 and 18 months after treatment
* Uterine size with MRI, before and 3 months after treatment.
* Aspect of the uterine cavity with hysteroscopy before and 3 months after treatment.
* Ovarian reserve with AMH dosage, and Antral follicular count before and 3 months after treatment.
* Volume and molecular pattern of the endometrium at the implantation window before and 3 months after treatment (optional).
* Treatment's adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 and ≤ 43 years old
* At least one interstitial fibroid more than 3 cm on MRIat MRI)
* with symptoms: genital bleeding, chronic pelvic pain or heaviness, anemia, or infertility > 1 year.
* With immediate desire to conceive
* without assisted reproductive indication: no tubal infertility, menstrual irregularities, hydrosalpinx, endometriosis, adenomyosis, or male infertility.
* Patient with health insurance, who can read and understand French and who has given written consent

Exclusion Criteria:

* Ongoing regnancy
* Emergency Situation
* Contraindication to surgery or uterine embolization: allergy to contrast medium , renal failure, immunodeficiency, contraindication to anesthesia, subserosal or submucosal pedunculated fibroids, fibroids with largest diameter inside of the uterine cavity

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Number of live birth in a year of fertility attempt | 18 months
  Women will be allowed to attempt fertility 6 months after treatment. Effective fertility attempts will be prospectively followed. Final fertility will be assessed one year later.

SECONDARY OUTCOMES:
number of adverse effects on fertility (ovarian reserve markers) | 18 months
number of adverse effects on fertility (state of the uterine cavity) | 18 months
number of adverse effects on fertility (state of the endometrium | 18 months
Improvement of symptoms related to fibroids With UFS-QoL questionnaires | 3 months
Improvement of symptoms related to fibroids With UFS-QoL questionnaires | 6 months
Improvement of symptoms related to fibroids With UFS-QoL questionnaires | 12 months
Improvement of symptoms related to fibroids With UFS-QoL questionnaires | 18 months
Quality of life With QSF questionnaires, a French version of the WHQ questionnaire | 3 months
Quality of life With QSF questionnaires, a French version of the WHQ questionnaire | 6 months
Quality of life With QSF questionnaires, a French version of the WHQ questionnaire | 12 months
Quality of life With QSF questionnaires, a French version of the WHQ questionnaire | 18 months
Number of adverse effects during pregnancy : Rate of Miscarriage | Until 30 months
Number of adverse effects during pregnancy : extra-uterine pregnancy | until 24 months
Number of adverse effects during pregnancy : small for gestational age | Until 30 months
Number of adverse effects during pregnancy : foetal death | Until 30 months
Number of adverse effects during pregnancy : uterine rupture | Until 30 months
Number of adverse effects during pregnancy : abnormal placental position and implantation | Until 30 months
Number of adverse effects during pregnancy : preterm delivery | Until 29 months
Number of adverse effects during pregnancy : delivery hemorrhagy | Until 30 months
number of adverse effects in the newborn | At day 3 of life
  Rate of small for gestational age, delivery presentation, health of newborn children (Apgar score, cord pH, admission in the neonatology service)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Torre, MD, PhD, Principal Investigator — Faculté de médecine de Montpellier-Nîmes, Université de Montpellier 1, France.; Arnaud Fauconnier, MD, PhD, Study Director — UFR des sciences de la santé Simone Veil, Université de Versailles Saint Quentin en Yvelines, France.
Locations (1):
- Département de Médecine de la Reproduction, Centre Hospitalier Régionnal Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta JK, Sinha A, Lumsden MA, Hickey M. Uterine artery embolization for symptomatic uterine fibroids. Cochrane Database Syst Rev. 2012 May 16;(5):CD005073. doi: 10.1002/14651858.CD005073.pub3. PMID 22592701
- [Background] Torre A, Paillusson B, Fain V, Labauge P, Pelage JP, Fauconnier A. Uterine artery embolization for severe symptomatic fibroids: effects on fertility and symptoms. Hum Reprod. 2014 Mar;29(3):490-501. doi: 10.1093/humrep/det459. Epub 2014 Jan 15. PMID 24430777
- [Background] Mara M, Maskova J, Fucikova Z, Kuzel D, Belsan T, Sosna O. Midterm clinical and first reproductive results of a randomized controlled trial comparing uterine fibroid embolization and myomectomy. Cardiovasc Intervent Radiol. 2008 Jan-Feb;31(1):73-85. doi: 10.1007/s00270-007-9195-2. Epub 2007 Oct 18. PMID 17943348